CLINICAL TRIAL: NCT04770389
Title: A Placebo-Controlled, Double-Blind, Randomized Phase 2 Study to Evaluate the Effect of Obicetrapib in Combination With Ezetimibe in Participants With Mild Dyslipidemia
Brief Title: Randomized Study of Obicetrapib in Combination With Ezetimibe
Acronym: OCEAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-303
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Dyslipidemias; High Cholesterol; Hypercholesterolemia
Keywords: obicetrapib; statin; LDL-C; cholesterol; atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe; Hypolipidemic Agents

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, Double-Blind, Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): placebo obicetrapib + placebo ezetimibe; once daily
  Interventions: Other: Placebo
- Combination therapy (Experimental): 5 mg obicetrapib + 10 mg ezetimibe; once daily
  Interventions: Drug: Obicetrapib 5mg; Drug: Ezetimibe 10mg
- Obicetrapib monotherapy (Experimental): 5 mg obicetrapib + placebo ezetimibe; once daily
  Interventions: Drug: Obicetrapib 5mg
- Ezetimibe monotherapy (Experimental): placebo obicetrapib + 10 mg ezetimibe; once daily
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Obicetrapib 5mg — tablet
  Other Names: CETP inhibitor
  Arms: Combination therapy; Obicetrapib monotherapy
Drug: Ezetimibe 10mg — tablet
  Other Names: Antihyperlipidemic
  Arms: Combination therapy; Ezetimibe monotherapy
Other: Placebo — tablet
  Arms: Placebo

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 2 study in participants with mild dyslipidemia to evaluate the efficacy, safety, and tolerability of obicetrapib and ezetimibe combination therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 2 study in participants with mild dyslipidemia to evaluate the efficacy, safety, and tolerability of obicetrapib and ezetimibe combination therapy. The screening period for this study will take up to 2 weeks. Following the screening period, eligible patients will be randomized to placebo, 5 mg obicetrapib + 10 mg ezetimibe; 5 mg obicetrapib + placebo ezetimibe; or placebo obicetrapib + 10 mg ezetimibe for an 8 week treatment period. After the treatment period, patients will continue for a 4 week safety follow-up and a 8 week PK follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study procedures, willingness to adhere to the study schedules and diet, and agreement to participate in the study by giving written informed consent prior to Screening procedures
* Men or women 18 to 70 years of age, inclusive
* Women may be enrolled if all 3 of the following criteria are met:
* They are not pregnant;
* They are not breastfeeding; and
* They do not plan on becoming pregnant during the study
* Women of childbearing potential must have a negative urine pregnancy test at the Screening Visit.
* Women of childbearing potential must agree to use an effective method of avoiding pregnancy from the Screening Visit to 90 days after the last visit. Men whose partners are of childbearing potential must agree to use an effective method of avoiding pregnancy from the Screening Visit to 90 days after the last visit.
* Fasting LDL-C levels >2.5 mmol/L (>100 mg/dL) and <4.5 mmol/L (<175 mg/dL) and TG levels <4.5 mmol/L (<400 mg/dL) (Visit 1) and
* Willingness to maintain a stable diet and physical activity level throughout the study

Exclusion Criteria:

* Body mass index >= 40 kg/m2
* Participation in another clinical study involving an investigational or marketed drug within 30 days prior to the Screening Visit
* Currently taking any lipid-altering therapy
* Any clinical manifestation of atherosclerotic CVD or any evidence of ischemic coronary disease present on the 12-lead ECG at the Screening Visit
* Diagnosis of type 1 or type 2 diabetes mellitus; or HbA1c >= 6.5% at the Screening visit if no prior diagnosis of diabetes mellitus
* Uncontrolled hypertension ie, sitting systolic blood pressure >160 mmHg and/or sitting diastolic blood pressure >90 mmHg taken as the average of triplicate measurements.

One retest will be allowed, at which point if the retest result is no longer exclusionary, the participant may be randomized

* Active muscle disease or persistent creatine kinase concentration >3 x the upper limit of normal (ULN). One retest will be allowed after 1 week to verify the result, at which point if the retest result is no longer exclusionary, the participant may be randomized
* History of torsades de pointes
* Estimated glomerular filtration rate <60 mL/min calculated using the Chronic Kidney Disease Epidemiology Collaboration equation
* Hepatic dysfunction as evidenced by any laboratory abnormality as follows: gamma- glutamyl transferase, alanine aminotransferase, or aspartate aminotransferase >2 x ULN, or total bilirubin >1.5 x ULN
* Anemia, defined as hemoglobin concentration <11 g/dL for males and hemoglobin concentration <9 g/dL for females
* History of malignancy within the past 5 years, with the exception of non-melanoma skin cancers
* Evidence of any other clinically significant non-cardiac disease or condition that, in the opinion of the Investigator, would preclude participation in the study
* Known ezetimibe or CETP inhibitor allergy or intolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Clinical Trials Research, Lincoln, California
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Juno Research, LLC - Medical Center Office, Houston, Texas
- Netherlands (6):
  - Huisartsen Praktijk A.M.N. Zijtregto, Rotterdam
  - Huisartsen Praktijk van Soerland, Rotterdam
  - Medisch Centrum Thomsonplein, The Hague
  - Huisartsen Praktijk Rambharose, The Hague
  - Huisartsen Praktijk Broekman, Zwijndrecht
  - Dokters van Nederhoven, Zwijndrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pirillo A, Catapano AL. The two faces of cholesteryl ester transfer protein inhibitors. Curr Opin Lipidol. 2025 Dec 1;36(6):318-325. doi: 10.1097/MOL.0000000000001017. Epub 2025 Oct 13. PMID 41190670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 234 participants were screened; out of 234, 112 participants were randomized. One participant in the ezetimibe 10 mg group was randomized in error and did not participate in the study or receive study drug
Period: Overall Study
Arm/Group | Placebo | Combination Therapy | Obicetrapib Monotherapy | Ezetimibe Monotherapy
Started | 28 | 27 | 28 | 29
Completed | 26 | 22 | 26 | 24
Not Completed | 2 | 5 | 2 | 5
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Failed attempt to draw blood | 1 | 0 | 0 | 0
Not completed — Left the country | 0 | 0 | 1 | 2
Not completed — Randomized in error and did not receive study drug | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Moved away from study site | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was revised from a 12-week treatment period to an 8-week treatment period in response to the global COVID-19 pandemic. Baseline Population is defined as all participants who received at least one dose of study drug and had a baseline value for LDL-C assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Combination Therapy | Obicetrapib Monotherapy | Ezetimibe Monotherapy | Total
Number analyzed (Participants) | 28 | 27 | 28 | 28 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.81) | 53.5 (11.43) | 59.1 (7.50) | 54.4 (9.55) | 55.4 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 14 | 14 | 60
  Male | 12 | 11 | 14 | 14 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 26 | 27 | 25 | 104
  Unknown or Not Reported | 2 | 1 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 4 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 24 | 22 | 23 | 24 | 93
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was calculated using the Friedewald Formula.
  milligrams per deciliter (mg/dL) | 136.8 (19.86) | 132.2 (27.48) | 127.5 (20.87) | 128.0 (22.33) | 131.13 (22.64)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [Friedewald]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 27
percent change from baseline | -45.63 (21.677) | -0.17 (12.682)
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -44.92, 95% CI 2-sided [-55.20 to -34.63], Standard Error of Mean 5.183

2. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [Friedewald]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 27
percent change from baseline | -51.95 [-77.9 to 3.1] | -1.40 [-20.9 to 33.6]
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -44.92, 95% CI 2-sided [-55.20 to -34.63], Standard Error of Mean 5.183

3. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [Friedewald]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 27 | 28
percent change from baseline | -43.55 (3.746) | 1.37 (3.604)
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -44.92, 95% CI 2-sided [-55.20 to -34.63], Standard Error of Mean 5.183

4. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [PUC]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 22
percent change from baseline | -44.38 (20.731) | -1.53 (15.105)
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -43.33, 95% CI 2-sided [-54.29 to -32.36], Standard Error of Mean 5.517

5. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [PUC]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 22
percent change from baseline | -51.40 [-69.6 to 8.1] | -2.00 [-24.5 to 35.9]
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -43.33, 95% CI 2-sided [-54.29 to -32.36], Standard Error of Mean 5.517

6. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo [PUC]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 22
percent change from baseline | -44.10 (3.813) | -0.78 (4.012)
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -43.33, 95% CI 2-sided [-54.29 to -32.36], Standard Error of Mean 5.517

7. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [Friedewald]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 25 | 27
percent change from baseline | -31.88 (18.860) | -0.17 (12.682)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -33.36, 95% CI 2-sided [-43.63 to -23.09], Standard Error of Mean 5.176

8. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [Friedewald]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 25 | 27
percent change from baseline | -34.40 [-57.0 to 23.8] | -1.40 [-20.9 to 33.6]
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -33.36, 95% CI 2-sided [-43.63 to -23.09], Standard Error of Mean 5.176

9. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [Friedewald]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 28 | 28
percent change from baseline | -31.99 (3.686) | 1.37 (3.604)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -33.36, 95% CI 2-sided [-43.63 to -23.09], Standard Error of Mean 5.176

10. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [PUC]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 25 | 22
percent change from baseline | -27.94 (18.914) | -1.53 (15.105)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -28.20, 95% CI 2-sided [-39.32 to -17.08], Standard Error of Mean 5.596

11. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [PUC]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 25 | 22
percent change from baseline | -30.10 [-56.7 to 19.1] | -2.00 [-24.5 to 35.9]
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -28.20, 95% CI 2-sided [-39.32 to -17.08], Standard Error of Mean 5.596

12. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo [PUC]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 25 | 22
percent change from baseline | -28.98 (3.802) | -0.78 (4.012)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean = -28.20, 95% CI 2-sided [-39.32 to -17.08], Standard Error of Mean 5.596

13. Secondary Outcome: Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: Mean percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 27
percent change from baseline | -31.62 (15.521) | -1.17 (11.692)
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -29.62, 95% CI 2-sided [-37.12 to -22.12], Standard Error of Mean 3.780

14. Secondary Outcome: Median Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: Median percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 24 | 27
percent change from baseline | -34.75 [-53.0 to 8.9] | -0.90 [-19.8 to 25.4]
Statistical Analysis 1: Comparison: Combination Therapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -29.62, 95% CI 2-sided [-37.12 to -22.12], Standard Error of Mean 3.780

15. Secondary Outcome: LS Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: LS Mean percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 27 | 28
percent change from baseline | -29.73 (2.730) | -0.11 (2.626)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -29.62, 95% CI 2-sided [-37.12 to -22.12], Standard Error of Mean 3.780

16. Secondary Outcome: Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo
Description: Mean percent change in Apo-B from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 26 | 27
percent change from baseline | -22.15 (13.356) | -1.17 (11.692)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -22.36, 95% CI 2-sided [-29.83 to -14.88], Standard Error of Mean 3.768

17. Secondary Outcome: Median Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo
Description: Median percent change in Apo-B from baseline to Day 57
Time Frame: 8 weeks
Population: The study was revised from a 12-week treatment period to an 8-week treatment period in response to the global COVID-19pandemic. Baseline Population is defined as all participants who received at least one dose of study drug and had a baselinevalue for LDL-C assessment.
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 26 | 27
percent change from baseline | -23.50 [-39.3 to 21.2] | -0.90 [-19.8 to 25.4]
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -22.36, 95% CI 2-sided [-29.83 to -14.88], Standard Error of Mean 3.768

18. Secondary Outcome: LS Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Placebo
Description: LS Mean percent change in Apo-B from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Placebo
Number analyzed (Participants) | 28 | 28
percent change from baseline | -22.46 (2.675) | -0.11 (2.626)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -22.36, 95% CI 2-sided [-29.83 to -14.88], Standard Error of Mean 3.768

19. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy [Friedewald]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 25
percent change from baseline | -45.63 (21.677) | -12.69 (21.316)
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -30.13, 95% CI 2-sided [-40.55 to -19.71], Standard Error of Mean 5.254

20. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy [Friedewald]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 25
percent change from baseline | -51.95 [-77.9 to 3.1] | -14.80 [-51.9 to 59.1]
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -30.13, 95% CI 2-sided [-40.55 to -19.71], Standard Error of Mean 5.254

21. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy [Friedewald]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 27 | 28
percent change from baseline | -43.55 (3.746) | -13.42 (3.675)
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -30.13, 95% CI 2-sided [-40.55 to -19.71], Standard Error of Mean 5.254

22. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Ezetimibe Monotherapy [Friedewald]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 25 | 25
percent change from baseline | -31.88 (18.860) | -12.69 (21.316)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Ezetimibe Monotherapy; Test type: Superiority; p = 0.0005, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -18.58, 95% CI 2-sided [-28.88 to -8.27], Standard Error of Mean 5.196

23. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Ezetimibe Monotherapy [Friedewald]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 25 | 25
percent change from baseline | -34.40 [-57.0 to 23.8] | -14.80 [-51.9 to 59.1]
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy vs Ezetimibe Monotherapy; Test type: Superiority; p = 0.0005, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -18.58, 95% CI 2-sided [-28.88 to -8.27], Standard Error of Mean 5.196

24. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Obicetrapib Monotherapy Compared to Ezetimibe Monotherapy [Friedewald]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C calculated using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Obicetrapib Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 28 | 28
percent change from baseline | -31.99 (3.686) | -13.42 (3.675)
Statistical Analysis 1: Comparison: Obicetrapib Monotherapy; Test type: Superiority; p = 0.0005, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -18.58, 95% CI 2-sided [-28.88 to -8.27], Standard Error of Mean 5.196

25. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [Friedewald]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C determined using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 25 | 27
percent change from baseline | -12.69 (21.316) | -0.17 (12.682)
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0051, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -14.79, 95% CI 2-sided [-25.03 to -4.54], Standard Error of Mean 5.165

26. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [Friedewald]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C calculated using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 25 | 27
percent change from baseline | -14.80 [-51.9 to 59.1] | -1.40 [-20.9 to 33.6]
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0051, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -14.79, 95% CI 2-sided [-25.03 to -4.54], Standard Error of Mean 5.165

27. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [Friedewald]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C calculated using the Friedewald formula
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 28 | 28
percent change from baseline | -13.42 (3.675) | 1.37 (3.604)
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0051, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -14.79, 95% CI 2-sided [-25.03 to -4.54], Standard Error of Mean 5.165

28. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [PUC]
Description: Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 23 | 22
percent change from baseline | -13.68 (19.573) | -1.53 (15.105)
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0245, ANCOVA; Least Squares (LS) Mean = -12.77, 95% CI 2-sided [-23.86 to -1.68], Standard Error of Mean 5.580

29. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [PUC]
Description: Median percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 23 | 22
percent change from baseline | -14.90 [-46.8 to 46.9] | -2.00 [-24.5 to 35.9]
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0245, ANCOVA; Least Squares (LS) Mean = -12.77, 95% CI 2-sided [-23.86 to -1.68], Standard Error of Mean 5.580

30. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 57: Ezetimibe Monotherapy Compared to Placebo [PUC]
Description: LS Mean percent change in LDL-C from baseline to Day 57; LDL-C measured using preparative ultracentrifugation (PUC)
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe Monotherapy | Placebo
Number analyzed (Participants) | 23 | 22
percent change from baseline | -13.55 (3.891) | -0.78 (4.012)
Statistical Analysis 1: Comparison: Ezetimibe Monotherapy vs Placebo; Test type: Superiority; p = 0.0245, ANCOVA; Least Squares (LS) Mean = -12.77, 95% CI 2-sided [-23.86 to -1.68], Standard Error of Mean 5.580

31. Secondary Outcome: Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy
Description: Mean percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 25
percent change from baseline | -31.62 (15.521) | -8.78 (14.445)
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -20.81, 95% CI 2-sided [-28.39 to -13.22], Standard Error of Mean 3.822

32. Secondary Outcome: Median Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy
Description: Median percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 25
percent change from baseline | -34.75 [-53.0 to 8.9] | -8.90 [-45.4 to 32.3]
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -20.81, 95% CI 2-sided [-28.39 to -13.22], Standard Error of Mean 3.822

33. Secondary Outcome: LS Mean Percent Change in Apolipoprotein-B (ApoB) From Baseline to Day 57: Obicetrapib in Combination With Ezetimibe Compared to Ezetimibe Monotherapy
Description: LS Mean Percent change in ApoB from baseline to Day 57
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Combination Therapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 27 | 28
percent change from baseline | -29.73 (2.730) | -8.92 (2.675)
Statistical Analysis 1: Comparison: Combination Therapy vs Ezetimibe Monotherapy; Test type: Superiority; p < 0.0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Mean = -20.81, 95% CI 2-sided [-28.39 to -13.22], Standard Error of Mean 3.822

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 16
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Combination Therapy | Obicetrapib Monotherapy | Ezetimibe Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/28 | 2/28
Other Adverse Events (participants affected / at risk) | 6/28 | 9/27 | 4/28 | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Combination Therapy (N=27) | Obicetrapib Monotherapy (N=28) | Ezetimibe Monotherapy (N=28)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Combination Therapy (N=27) | Obicetrapib Monotherapy (N=28) | Ezetimibe Monotherapy (N=28)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04770389/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04770389/SAP_001.pdf